CLINICAL TRIAL: NCT00418002
Title: A Randomized, Double-Blind, Ascending Dose, Placebo-Controlled Single Dose Study in Non-Smoking Healthy Elderly Subjects Interleaved With a 2-Week Multiple Once Daily Dose Study to Explore Safety, Tolerability, Pharmacokinetics and Cognitive Effects After Oral Administration of AQW051
Brief Title: Safety and Tolerability of AQW051 in Elderly Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAQW051A2102
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Single-rising dose , multiple rising dose, elderly, cognitive, , pharmacokinetic, impairment.; Healthy elderly male and female subjects
MeSH Terms: interventions — 3-(6-p-tolylpyridin-3-yloxy)-1-azabicyclo(2.2.2)octane

INTERVENTIONS:
Drug: AQW051

SUMMARY:
The purpose of this study is to assess safety and tolerability of AQW051 administered in single and multiple doses to elderly healthy volunteers. In addition, pharmacokinetic effects will be assessed and the possible effects on cognition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and postmenopausal female subjects between 60 to 80 years of age and in good health as determined by past medical history.
* Postmenopausal women must have no regular menstrual bleeding for at least 1 year prior to inclusion.
* Male subjects must be using a double-barrier local contraception.
* Body mass index must be within the range of 18 to 33. Subjects must weigh at least 50 kg to participate in this study.
* The regular intake of concomitant drugs including thyroxine, paracetamol, low dose non-steroidal anti-inflammatory drugs, lipid lowering drugs, vitamins and dietary supplements without caffeine and nicotinic acid, and hormone replacement therapy is allowed, if on stable treatment for at least 3 months. Intake of nutritional supplements (e.g. omega-3, vitamins, minerals, cod-liver oil) is allowed.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent.

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months).
* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (e.g. herbal supplements) within 2 weeks prior to study start except noted previously
* Use of any central nervous system active drug and anticholinergic drugs during the previous 3 months and use of any drug or treatment known to cause major organ system toxicity during the previous 3 months is prohibited.
* A past personal or close family medical history of clinically significant cardiac abnormalities.
* Current diagnosis of cardiac arrhythmia derived from ECG and/or Holter ECG.
* Current diagnosis of cardiovascular disease.
* Current diagnosis or history of autonomic dysfunction (e.g. history of fainting, orthostatic hypotension, sinus arrhythmia).
* History of Acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease) Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis) Known hypersensitivity or severe adverse event to darifenacin or similar drugs Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize participation in the study Immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result. Drug or alcohol abuse within the 12 months prior to dosing.
* Diagnosis of cognitive impairment (Mini Mental State Exam < 27).
* History or current diagnosis of a cerebrovascular disease (e.g., stroke, transient ischemic attacks, aneurysms).
* Current DSM-IV diagnosis of major depression and/or any other DSM-IV Axis 1 diagnosis that may interfere with the evaluation of the patient's response to study medication, including other primary neurodegenerative dementia, schizophrenia, or bipolar disorder.
* History or current diagnosis of an active, uncontrolled seizure disorder.
* History of head injury or any other neurological disorder.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Safety and tolerability.

SECONDARY OUTCOMES:
Pharmacokinetics at the end of the study.
Effect of AQW051 on cognition as assessed by a computerized cognitive test battery.
To assess a potential food effect on pharmacokinetics of AQW051.
To explore the drug abuse liability potential of AQW051.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Horsham, United Kingdom